CLINICAL TRIAL: NCT00005461
Title: Epidemiology of Symptom Perception in Childhood Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4905; R01HL045157 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To investigate the determinants of valid symptom perception in childhood asthma and the relation of symptom perception to asthma morbidity.

DETAILED DESCRIPTION:
BACKGROUND:

The treatment of childhood asthma increasingly entails self-management as an important factor in influencing the course of the disease. The study identified subgroups of children who were at increased risk of misinterpreting, and thus mismanaging, their pulmonary function. Identification of the characteristics of these high risk children formed the basis for subsequent development of an intervention program to improve symptom self-perception, thereby enhancing the children's ability to participate effectively in self-management of their asthma.

DESIGN NARRATIVE:

The specific hypotheses tested in the cross-sectional prevalence study were: 1) greater validity of self-perceived symptoms was associated with less functional morbidity from asthma; 2) specific psychological and asthma-related determinants affected the sensitivity and specificity of symptom perception in children with asthma; 3) perception of respiratory symptoms was a measurable characteristic that could be evaluated in terms of reliability and validity; 4) perceptual accuracy in a natural or clinical setting was significantly related to perceptual ability measured in a laboratory.

Investigation of these objectives used a study of validity of self-perception of symptoms in relation to clinical status. Children aged 8-15 made subjective estimates of their asthma severity immediately prior to pulmonary function testing at multiple times while they lived either at a summer camp for children with asthma or a long-term asthma treatment center. The correspondence between subjective and objective measures of pulmonary function in the clinical environment were compared with results obtained in a laboratory using threshold detection of added resistive loads. The sensitivity and specificity of asthmatic children's self-assessment of symptom state were quantified and related retrospectively to risk of functional morbidity. Cognitive abilities, anxiety level, tendency toward repression, locus of control, and familial factors were investigated regarding their role as determinants of sensitivity and specificity of symptom self-perception as a measure of pulmonary function. The stability of individual patterns of self-perception were studied longitudinally with annual repeated evaluations among those children who returned to camp or were rehospitalized.

The study with its three-component research plan was renewed in fiscal year 1997. Component 1 strengthened understanding of the psychologic and physiologic correlates of perceptual ability. A positive association was expected between perceptual accuracy and a) intelligence; b) attention; c) symptom focus; d) systemic steroid use; and e) predominantly large airway or mixed airway involvement. Component 2 explored the relationship between chemosensitivity and resistive-load perception in high risk pediatric asthma patients. It was hypothesized that, compared to other asthmatics and controls, adolescents who had near fatal asthma attacks a) had higher thresholds for detecting resistive loads; b) had a decreased response to progressive isocapneic hypoxia; and c) had a smaller increase in respiratory drive during progressive hypercapnia. Component 3 characterized the family and self-management patterns moderating variables between perception and morbidity. It was hypothesized that a) symptom perception interacted with family asthma management in relation to asthma morbidity b) poor symptom perception was associated with worse medication compliance; and c) better family functioning was related to better perception and lower functional morbidity. Methodologic approaches included a naturalistic clinical accuracy protocol; laboratory studies using a computerized resistive-loading apparatus to determine perceptual thresholds; a chemosensitivity protocol investigating drive; family assessment interviews, and computerized metered dose inhaler technology to assess compliance with asthma medications.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-04; Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Fritz — Rhode Island Hospital

REFERENCES:
- [Background] Fritz GK, Yeung A, Wamboldt MZ, Spirito A, McQuaid EL, Klein R, Seifer R. Conceptual and methodologic issues in quantifying perceptual accuracy in childhood asthma. J Pediatr Psychol. 1996 Apr;21(2):153-73. doi: 10.1093/jpepsy/21.2.153. PMID 8920151
- [Background] Fritz GK, McQuaid EL, Spirito A, Klein RB. Symptom perception in pediatric asthma: relationship to functional morbidity and psychological factors. J Am Acad Child Adolesc Psychiatry. 1996 Aug;35(8):1033-41. doi: 10.1097/00004583-199608000-00014. PMID 8755800
- [Background] Klein RB, Fritz GK, Yeung A, McQuaid EL, Mansell A. Spirometric patterns in childhood asthma: peak flow compared with other indices. Pediatr Pulmonol. 1995 Dec;20(6):372-9. doi: 10.1002/ppul.1950200607. PMID 8649917
- [Background] Fritz G, Spirito A, Yeung A, Klein R, Freedman E. A pictorial visual analog scale for rating severity of childhood asthma episodes. J Asthma. 1994;31(6):473-8. doi: 10.3109/02770909409089489. PMID 7961324
- [Background] Fritz GK, Yeung A, Taitel MS. Symptom perception and self-management in childhood asthma. Curr Opin Pediatr. 1994 Aug;6(4):423-7. doi: 10.1097/00008480-199408000-00012. PMID 7951663
- [Background] Fritz GK, McQuaid EL, Nassau JH, Klein RB, Mansell A. Thresholds of resistive load detection in children with asthma. Pediatr Pulmonol. 1999 Oct;28(4):271-6. doi: 10.1002/(sici)1099-0496(199910)28:43.0.co;2-c. PMID 10497376
- [Background] Gavin LA, Wamboldt MZ, Sorokin N, Levy SY, Wamboldt FS. Treatment alliance and its association with family functioning, adherence, and medical outcome in adolescents with severe, chronic asthma. J Pediatr Psychol. 1999 Aug;24(4):355-65. doi: 10.1093/jpepsy/24.4.355. PMID 10431501
- [Background] Frankel K, Wamboldt MZ. Chronic childhood illness and maternal mental health--why should we care? J Asthma. 1998;35(8):621-30. doi: 10.3109/02770909809048964. PMID 9860082
- [Background] Wamboldt MZ, Schmitz S, Mrazek D. Genetic association between atopy and behavioral symptoms in middle childhood. J Child Psychol Psychiatry. 1998 Oct;39(7):1007-16. PMID 9804033
- [Background] Wamboldt MZ, Fritz G, Mansell A, McQuaid EL, Klein RB. Relationship of asthma severity and psychological problems in children. J Am Acad Child Adolesc Psychiatry. 1998 Sep;37(9):943-50. doi: 10.1097/00004583-199809000-00014. PMID 9735613
- [Background] Wamboldt MZ, Yancey AG Jr, Roesler TA. Cardiovascular effects of tricyclic antidepressants in childhood asthma: a case series and review. J Child Adolesc Psychopharmacol. 1997 Spring;7(1):45-64. doi: 10.1089/cap.1997.7.45. PMID 9192541
- [Background] Bender B, Wamboldt FS, O'Connor SL, Rand C, Szefler S, Milgrom H, Wamboldt MZ. Measurement of children's asthma medication adherence by self report, mother report, canister weight, and Doser CT. Ann Allergy Asthma Immunol. 2000 Nov;85(5):416-21. doi: 10.1016/s1081-1206(10)62557-4. PMID 11101187
- [Background] Wamboldt FS, O'Connor SL, Wamboldt MZ, Gavin LA, Klinnert MD. The five minute speech sample in children with asthma: deconstructing the construct of expressed emotion. J Child Psychol Psychiatry. 2000 Oct;41(7):887-98. PMID 11079431
- [Background] Gabriels RL, Wamboldt MZ, McCormick DR, Adams TL, McTaggart SR. Children's illness drawings and asthma symptom awareness. J Asthma. 2000;37(7):565-74. doi: 10.3109/02770900009090811. PMID 11059523
- [Background] Wamboldt MZ, Wamboldt FS. Role of the family in the onset and outcome of childhood disorders: selected research findings. J Am Acad Child Adolesc Psychiatry. 2000 Oct;39(10):1212-9. doi: 10.1097/00004583-200010000-00006. PMID 11026173
- [Background] McQuaid EL, Fritz GK, Nassau JH, Lilly MK, Mansell A, Klein RB. Stress and airway resistance in children with asthma. J Psychosom Res. 2000 Oct;49(4):239-45. doi: 10.1016/s0022-3999(00)00173-2. PMID 11119780
- [Background] Wamboldt FS, Price MR, Hume LA, Gavin LA, Wamboldt MZ, Klinnert MD. Reliability and validity of a system for coding asthma outcomes from medical records. J Asthma. 2002 Jun;39(4):299-305. doi: 10.1081/jas-120002286. PMID 12095179
- [Background] Wamboldt FS, Ho J, Milgrom H, Wamboldt MZ, Sanders B, Szefler SJ, Bender BG. Prevalence and correlates of household exposures to tobacco smoke and pets in children with asthma. J Pediatr. 2002 Jul;141(1):109-15. doi: 10.1067/mpd.2002.125490. PMID 12091860
- [Background] Wamboldt MZ, Wamboldt FS, Gavin L, McTaggart AS. A parent-child relationship scale derived from the child and adolescent psychiatric assessment (CAPA). J Am Acad Child Adolesc Psychiatry. 2001 Aug;40(8):945-53. doi: 10.1097/00004583-200108000-00017. PMID 11501695
- [Background] Millikan E, Wamboldt MZ, Bihun JT. Perceptions of the family, personality characteristics, and adolescent internalizing symptoms. J Am Acad Child Adolesc Psychiatry. 2002 Dec;41(12):1486-94. doi: 10.1097/00004583-200212000-00021. PMID 12447036
- [Background] Wamboldt MZ, Laudenslager M, Wamboldt FS, Kelsay K, Hewitt J. Adolescents with atopic disorders have an attenuated cortisol response to laboratory stress. J Allergy Clin Immunol. 2003 Mar;111(3):509-14. doi: 10.1067/mai.2003.140. PMID 12642830
- [Background] Bihun JT, Wamboldt MZ, Gavin LA, Wamboldt FS. Can the Family Assessment Device (FAD) be used with school aged children? Fam Process. 2002 Winter;41(4):723-31. doi: 10.1111/j.1545-5300.2002.00723.x. PMID 12613127
- [Background] Klein RB, Walders N, McQuaid EL, Adams S, Yaros D, Fritz GK. The Asthma Risk Grid: clinical interpretation of symptom perception. Allergy Asthma Proc. 2004 Jan-Feb;25(1):1-6. PMID 15055553